CLINICAL TRIAL: NCT00953940
Title: Prevention of Perioperative Acute Renal Failure in Abdominal Surgery
Brief Title: Prevention of Perioperative Acute Renal Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: An external board recommended to close the study for futility after the interin analysis
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Fernando Liaño García, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Nefrane001; NºEudra CT: 2005-004755-35
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2009-08

CONDITIONS: Abdominal Surgery
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isotonic saline (Experimental): Isotonic saline
  Interventions: Drug: Isotonic saline
- No treatment (No Intervention): Habitual therapy

INTERVENTIONS:
Drug: Isotonic saline — Isotonic saline administrated i.v at 1.5 ml/Kg/h , 8 to 12 h before surgery
  Arms: Isotonic saline

SUMMARY:
The purpose of this study is to measure the acute renal dysfunction on the first, second, seventh and twentieth days.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are undergoing elective abdominal surgery after appropriate information of the study, and its possible risks that may arise therefrom and that at any time to refuse their cooperation, give a written consent to participate in the study.
* Patients who at the time of the interview have an ASA between 2 and 4.
* Patients with chronic kidney failure mild moderate (serum creatinine between 1.5 and 3.0 mg / dl) can be included.

Exclusion Criteria:

* Chronic kidney diseases with serum creatinine higher than 3.0 mg /DL
* Laparoscopic abdominal surgery
* ASA 1 and ASA 5 patients.
* Patients with cardiac insufficiency, ascites and respiratory insufficiency
* Diastolic hypertension > 100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-06; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Serum creatinine in the first, second, seventh and twenty after surgery in patients undergoing elective abdominal surgery. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Fernando Liaño, MD PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Ramon y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Serrano AB, Candela-Toha AM, Zamora J, Vera J, Muriel A, Del Rey JM, Liano F. Preoperative hydration with 0.9% normal saline to prevent acute kidney injury after major elective open abdominal surgery: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jun;33(6):436-43. doi: 10.1097/EJA.0000000000000421. PMID 26825017